CLINICAL TRIAL: NCT01016847
Title: A Randomized, Double-Blind, Placebo-Controlled, Cross-over Study to Evaluate the Effect of the Leukotriene Antagonist (Singulair©) Plus Moderate Dose Beclomethasone Compared to High Dose Beclomethasone in Obese Subjects With Moderate Persistent Asthma
Brief Title: Moderate to Persistent Asthma in the Obese Subject
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to enroll enough study subjects. Study has been terminated
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: Pro00018748
Record Dates: First submitted 2009-10-19; First posted 2009-11-20 (Estimated); Results first posted 2014-11-17 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2012-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — montelukast; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- leukotriene receptor antagonist (LTRA) montelukast (Active Comparator): Montelukast (LTRA) administered with moderate dose of inhaled steroid
  Interventions: Drug: Montelukast
- Sugar Pill (Placebo Comparator): High dose of inhaled steroid administered with sugar pill
  Interventions: Other: Sugar pill

INTERVENTIONS:
Drug: Montelukast — 10 mg Q day
  Arms: leukotriene receptor antagonist (LTRA) montelukast
Other: Sugar pill — Sugar pill that looks like Montelukast that will be given Q day
  Arms: Sugar Pill

SUMMARY:
Obesity is associated with increased airway inflammation and asthma severity that results in suboptimal control of asthma despite therapy with high dose inhaled corticosteroids (ICS). The investigators suggested that the addition of Singular (montelukast)[LTRA] to moderate doses of inhaled corticosteroids will improve asthma control. This cross over study will be treat subjects with moderate dose ICS/LTRA for 12 weeks and high dose ICS with placebo for 12 weeks.

DETAILED DESCRIPTION:
Subjects will enter the 2-week run-in period after meeting eligibility criteria at the screening visit (visit 1). During run-in subjects will have all usual asthma medications discontinued and will be placed on inhaled corticosteroids at moderate doses and leukotriene receptor antagonists will be withdrawn (LTRA wash-out). Subjects will be monitored to rule out any acute infection or symptoms consistent with an exacerbation. The run-in period will be used to assess subject compliance and understanding of study related procedures. Following the run-in, to be eligible for the randomization subjects must have an ACQ score >1.25 on the Juniper Asthma Control Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* moderate persistent asthma as defined daily symptoms, nocturnal awakenings >1 time/week but not daily, daily short-acting beta agonist usage
* pre-bronchodilator Force expiratory volume (FEV1)>55% but <90%.
* Subjects must be on controller therapy for asthma with ICS for at least one month prior to enrollment.
* methacholine testing that causes a drop in the FEV1 of 20% (8mg/ml off ICS or 16mg/ml) on ICS within 6 months prior to entry
* physician diagnosis of asthma for at least one year prior to study enrollment.
* Obesity defined as BMI greater than 30.
* subjects must have an Asthma Control Questionnaire (ACQ) score >1.25 on the Juniper Asthma Control Questionnaire (indicating poor asthma control),
* require daily medications for asthma and be compliant with study related medications.

Exclusion Criteria:

* Subjects must not have been intubated in the last 5 years or unstable asthma symptoms resulting in significant loss or work or school
* upper or lower respiratory tract infection within 1 month of the study
* use of antibiotics within 4 weeks of the study
* use of oral glucocorticoids within 4 weeks
* use of theophylline
* smoking history greater than 10 pack years or any cigarette use within the past two years
* significant non-asthma pulmonary disease or other medical problems
* Subjects planning to undergo gastric bypass surgery within 4 months of the enrollment date will be excluded since weight loss is a potential confounder of asthma control
* Pregnant women will also be excluded

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke Asthma Allergy and Airway Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 38 subjects enrolled in study. Of the 38 subjects 10 were screen failures, and 25 were withdrawn during the 2 week run-in period.
Period: Overall Study
Arm/Group | Leukotriene Receptor Antagonist (LTRA) Montelukast | Sugar Pill
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Leukotriene Receptor Antagonist (LTRA) Montelukast | Sugar Pill | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Determine the Effect of Montelukast / Moderate Dose ICS Versus High Dose ICS on Asthma Control as Measured by the Asthma Control Questionnaire.
Time Frame: Baseline/randomization to week 16
Population: Due to insufficient accrual, data analysis was not performed.
Arm/Group | Leukotriene Receptor Antagonist (LTRA) Montelukast | Sugar Pill
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Serum Adiponectin, Leptin, Tumor Necrosis Alpha (TNF-α) and Interleukin 6 (IL6) Levels
Time Frame: Baseline/randomization to week 16
Population: Due to insufficient accrual, data analysis was not performed.
Arm/Group | Leukotriene Receptor Antagonist (LTRA) Montelukast | Sugar Pill
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Post Bronchodilator Forced Expiratory Volume in 1 Second (FEV1)
Time Frame: Baseline/randomization to week 16
Population: Due to insufficient accrual, data analysis was not performed.
Arm/Group | Leukotriene Receptor Antagonist (LTRA) Montelukast | Sugar Pill
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Trends in Asthma Control Questionnaire (ACQ ACTQ) Scores Over Duration of the Study
Time Frame: Baseline/randomization to week 16
Population: Due to insufficient accrual, data analysis was not performed.
Arm/Group | Leukotriene Receptor Antagonist (LTRA) Montelukast | Sugar Pill
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Asthma Exacerbation
Description: Asthma exacerbation is defined as the development of an increase in asthma symptoms which results in an increase in the use of asthma medications (typically inhaled corticosteroids and/or parenteral corticosteroids) or the addition of another new asthma medication or antibiotics.
Time Frame: Baseline/randomization to week 16
Population: Due to insufficient accrual, data analysis was not performed.
Arm/Group | Leukotriene Receptor Antagonist (LTRA) Montelukast | Sugar Pill
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Sputum Cell Counts and Differentials
Time Frame: Baseline/randomization to week 16
Population: Due to insufficient accrual, data analysis was not performed.
Arm/Group | Leukotriene Receptor Antagonist (LTRA) Montelukast | Sugar Pill
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline to week 16
Arm/Group | Leukotriene Receptor Antagonist (LTRA) Montelukast | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 0/2

LIMITATIONS AND CAVEATS:
Early terminiation due to poor enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No